CLINICAL TRIAL: NCT05691140
Title: Prevention of Postpartum Anxiety in High-Risk Women: A Proof-of-Concept Randomized Clinical Trial
Brief Title: Prevention of Postpartum Anxiety in High-Risk Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Sheryl Green, Clinical Psychologist, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13902
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Postpartum Anxiety
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioural Therapy (Experimental)
  Interventions: Other: Cognitive Behavioural Therapy
- Treatment as Usual (No Intervention)

INTERVENTIONS:
Other: Cognitive Behavioural Therapy — Cognitive Behavioural Therapy targeting Intolerance of Uncertainty
  Arms: Cognitive Behavioural Therapy

SUMMARY:
The primary aim of this study is to evaluate whether a CBT group designed to target IU (CBT-IU) in pregnant women with heightened levels of IU, prevents postpartum anxiety. The investigators hypothesize that women with clinically significant IU during pregnancy will exhibit both significant reductions in IU, as well as a decrease in anxiety symptoms postpartum, compared to a treatment as usual control group. The secondary aim of this study is to evaluate whether CBT-IU significantly improves and/or prevents depression symptoms, worry symptom severity, and difficulties with emotion regulation. The investigators hypothesize that CBT-IU will lead to significant improvements in symptom severity compared to the treatment as usual control group.

DETAILED DESCRIPTION:
Anxiety disorders are a serious mental health concern, affecting as many as 15-24% of women during the perinatal period. Despite the high prevalence of anxiety during the perinatal period and its associated impact, fewer than 15% of women receive treatment often due to difficulties in timely and accurate symptom detection. Our group conducted a longitudinal study that investigated the psychosocial and biological risk factors of postpartum anxiety worsening in a sample of high-risk pregnant women with pre-existing anxiety and depressive disorders. In this study, intolerance of uncertainty (IU) was identified as the strongest predictor. IU is a cardinal trait of anxiety and has been implicated in predicting treatment response in non-perinatal populations. However, despite the relevance of IU in anxiety disorders, our study was the first to assess IU in the perinatal population. As improving symptom detection through identification of significant risk factors, such as IU, can aid in the development of preventative and treatment measures, our group recently validated the Intolerance of Uncertainty Scale (IUS) in a perinatal population for the detection of anxiety disorders. In this study of 198 perinatal women, the IUS demonstrated excellent internal consistency and an optimal clinical cut-off score of 64 or greater was established, yielding a sensitivity of 89%. The IUS also demonstrated very good positive (79%) and negative (80%) predictive values. These findings suggest that the IUS represents a clinically useful screening tool to be used as an aid for the early and accurate detection of anxiety disorders during the perinatal period. Cognitive Behavioural Therapy (CBT) is considered a first-line treatment for perinatal anxiety disorders and CBT programs targeting IU have revealed promising findings in non-perinatal populations.It is therefore imperative to investigate whether a treatment program specifically designed to target IU during pregnancy can prevent postpartum anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (up to 30 weeks pregnant to allow for completion of the CBT-IU protocol before child delivery)
* 18 years or older
* Baseline score of ≥64 on the IUS (Furtado et al., 2021)
* No psychotropic medication or, if taking medication, no change in dose or type for a minimum of 6 weeks prior to baseline
* No concurrent psychological treatment
* Fluent in English and able to consent for treatment
* Located in Ontario, Canada

Exclusion Criteria:

* A current diagnosed DSM-5 anxiety disorder, as assessed by the Mini International Neuropsychiatric Interview (version 7.0.2)
* Active suicidal ideation
* Current psychosis or substance use disorder
* For those enrolled on a stable dosage of a psychotropic medication, if a change in medication is required during the psychological therapy trial, the participant will continue with the therapy but will be excluded from the analysis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with principal anxiety disorder (as per DSM-5) | 6-12 weeks postpartum
  Postpartum anxiety prevention will be defined as whether participants meet provisional DSM-5 diagnostic criteria for an anxiety disorder at the post-treatment assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl M Green, PhD, CPsych, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dennis CL, Falah-Hassani K, Shiri R. Prevalence of antenatal and postnatal anxiety: systematic review and meta-analysis. Br J Psychiatry. 2017 May;210(5):315-323. doi: 10.1192/bjp.bp.116.187179. Epub 2017 Mar 16. PMID 28302701
- [Background] Furtado M, Frey BN, Green SM. Validation of the intolerance of uncertainty scale as a screening tool for perinatal anxiety. BMC Pregnancy Childbirth. 2021 Dec 14;21(1):829. doi: 10.1186/s12884-021-04296-1. PMID 34903196
- [Background] Smith MV, Shao L, Howell H, Wang H, Poschman K, Yonkers KA. Success of mental health referral among pregnant and postpartum women with psychiatric distress. Gen Hosp Psychiatry. 2009 Mar-Apr;31(2):155-62. doi: 10.1016/j.genhosppsych.2008.10.002. Epub 2008 Dec 3. PMID 19269536
- [Background] Furtado M, Van Lieshout RJ, Van Ameringen M, Green SM, Frey BN. Biological and psychosocial predictors of anxiety worsening in the postpartum period: A longitudinal study. J Affect Disord. 2019 May 1;250:218-225. doi: 10.1016/j.jad.2019.02.064. Epub 2019 Mar 1. PMID 30870771
- [Background] Dugas MJ, Ladouceur R. Treatment of GAD. Targeting intolerance of uncertainty in two types of worry. Behav Modif. 2000 Oct;24(5):635-57. doi: 10.1177/0145445500245002. PMID 11036732
- [Background] van der Heiden C, Muris P, van der Molen HT. Randomized controlled trial on the effectiveness of metacognitive therapy and intolerance-of-uncertainty therapy for generalized anxiety disorder. Behav Res Ther. 2012 Feb;50(2):100-9. doi: 10.1016/j.brat.2011.12.005. Epub 2011 Dec 21. PMID 22222208
- [Derived] Furtado M, Frey BN, Inness BE, McCabe RE, Green SM. Targeting Intolerance of Uncertainty During Pregnancy: A Randomized Controlled Trial to Prevent Postpartum Anxiety Disorders. J Clin Psychiatry. 2025 Nov 5;87(1):25m15979. doi: 10.4088/JCP.25m15979. PMID 41190888
- [Derived] Furtado M, Frey BN, Inness BE, McCabe RE, Green SM. Cognitive behavioural therapy for intolerance of uncertainty: A study protocol for the prevention of postpartum anxiety. J Reprod Infant Psychol. 2025 Apr 29:1-20. doi: 10.1080/02646838.2025.2495928. Online ahead of print. PMID 40297898